CLINICAL TRIAL: NCT04326543
Title: Association Between Temperament Dimensions and Awakening Salivary Cortisol Levels in Children and Adolescents With Attention Deficit Hyperactivity/Impulsivity Disorder (ADHD)
Brief Title: Temperament Dimensions and Awakening Salivary Cortisol Levels in ADHD.
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, ALESSANDRA CARTA, Medical Doctor, PhD student, Università degli Studi di Sassari
Other Study IDs: 2472/CE
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva sample to tests awakening cortisol levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADHD and typically developing controls: 120 subject: 53 with an ADHD clinical diagnosis and 57 typically developing controls aged between 3 and 16 years old.
  Interventions: Diagnostic Test: Swanson, Noolan and Phelham - IV edition (SNAP-IV); Conners' Parent Rating Scales (CPRS)

INTERVENTIONS:
Diagnostic Test: Swanson, Noolan and Phelham - IV edition (SNAP-IV); Conners' Parent Rating Scales (CPRS) — * Ratings on the Swanson, Nolan and Pelham Evaluation Scale - IV (Bussing et al., 2008), were assessed during baseline visit for participants at the time of research assessment, to exclude the presence of ADHD symptoms in the healthy subjects. This scale is composed of 26 items for ADHD symptoms and ODD and was administered at baseline and at follow-up visit.
  * Temperament assessment: we used the Mary Rothbart's Temperament Questionnaire, a caregivers' report measure designed to provide a detailed assessment of temperament.
  * ADHD Rating scales: the Long Version of Conners' Parent Rating Scale (Conners et al., 1998) was used to quantify ADHD comorbidity symptoms, as ODD and Anxiety traits, in the children and adolescents with ADHD.
  * Salivary cortisol: Sampling was performed during one ordinary weekday between 7 and 8 o'clock, within 60' after nocturnal awakening.
  Other Names: Rothbart Temperament questionnaires

SUMMARY:
To analyze heterogeneity in ADHD experts in last decade advised to look beyond the lists of existing symptoms towards phenotypic measures that can be represented dimensionally and have well-theorized relationships with neurobiological systems, (Sonuga-Barke & Halperin, 2010; Insel et al, 2010; Fair D, Bathula D, Nikolas M, Nigg JT, 2012; Georgiades S, Szatmari P, Boyle M, 2013; Sanislow CA, Pine DS, Quinn KJ, et al, 2013). This is the nucleus of RDoC aims because children and adolescents with ADHD can be characterized in terms of several features that are best represented as dimensions and have well-theorized relationships to biological systems (Cuthbert & Insel, 2013).

DETAILED DESCRIPTION:
Recently evidence suggests that measures of child temperament may predict ADHD symptoms (Einziger et al., 2018). Temperament is a characteristic of personality (Buss & Plomin, 1984; Crowell, 2016) and refers to individual, neurobiologically-based difference in reactivity, self-regulation and cognition (Eisenberg, 2012).

It has been previously emphasized (Nigg J., 2016), that Hypotalamic-Pituitary-Adrenal (HPA) axis, through the cortisol hormone, may represent a powerful biological measure of behavioural self-regulatory systems, activity level, cognition, temperament (Stadler et al, 2011; Martel et al., 2009; Sonuga-Barke, 2005) and arousal (Snoek, Van Goozen, Matthys, Buitelaar, & Engeland, 2004). Cortisol is released from the surrenal gland by means of the HPA axis activation, in response to catecholaminergic neurotransmitters (Ulrich-Lai & Herman, 2009). Cortisol is involved in the regulation of a wide range of body functions, including emotion processing (Skosnik, Chatterton, Swisher, & Park, 2000), awakening (Fries, Dettenborn, & Kirschbaum, 2009) and stress responses (Chrousos, Kino, & Charmandari, 2009).

Both cortisol and temperament may share self-response regulatory processes (Martel et al., 2008; Nigg, 2016; Ulrich-Lai & Herman, 2009), and one study on 70 healthy pre-schoolers indicates that children with SE temperament has higher morning salivary cortisol levels during their first week of a new primary school year (Davis, Donzella, Krueger, & Gunnar, 1999), hypothesized as a stress-induced effect.

To date, no studies have been conducted to study heterogeneity starting from the self-response regulatory processes between temperament and cortisol in children and adolescents with ADHD.

As for clinical application of HPA-axis and cortisol level in ADHD diagnosis and dimension, available studies are, as yet, either inconsistent (Bonvicini, Faraone, & Scassellati, 2016; Freitag et al, 2009, Corominas et al, 2012) or suggestive, but not significant, upon dimensional stratification of ADHD symptoms (Pinto et al., 2016).

The aims of this study to contribute to the issue of clinical heterogeneity of ADHD, analysing whether ADHD symptoms and co-morbidity traits simultaneously link to both cortisol level and temperament dimensions, as biomarkers of arousal and inhibited behaviour. To pursue our aim we formulated five specific research questions: i) Do temperament dimensions and awakening cortisol level differ between children and adolescents with ADHD and TDC? ii) Do temperament dimensions and awakening cortisol levels correlate with dimension of ADHD core symptoms? iii) Does awakening cortisol level associate with any of the three-temperament dimension? iv) Do parent ratings of the oppositional and defiant traits and anxiety traits affect the association between temperament dimensions and cortisol levels with ADHD core symptoms in the ADHD group?

ELIGIBILITY:
Inclusion Criteria:

1. ADHD group:

   * The assessment was completed as part of their routine psychiatric assessment using unstructured interview, screening of ADHD and other psychiatric symptoms through parent questionnaires, and direct observation with the participants, which led to a DSM-5-based diagnosis of ADHD;
   * Signed informed consent from parents or legal guardian and/or assent for youth aged >12 y/o.
2. TDY (Typically Developing Control) - group:

   * Signed informed consent from parents or legal guardian and/or assent for youth aged >12 y/o;
   * TDY were recruited from pre-school, primary and secondary schools in the local catchment area.
   * Assessment of the TDY was carried out by a clinician in schools through an unstructured interview with the parents and teachers.

Exclusion Criteria:

1. ADHD group:

   * Not signed informed consent from parents or legal guardian and/or assent for youth aged >12 y/o;
   * IQ below 70;
   * neurological and other psychiatric disorders;
   * genetic and/or medical conditions mimicking ADHD symptoms;
   * treatment with psychotropic medications other than ADHD medications;
   * TDY were also excluded if they presented with any learning or behavioural difficulties as reported in the parent and teacher interviews, as well as mild, moderate or severe symptoms of ADHD in the clinician-led rating scale.
2. TDY (Typically Developing Control) - group:

   * Not signed informed consent from parents or legal guardian and/or assent for youth aged >12 y/o;
   * IQ below 70;
   * neurological and other psychiatric disorders;
   * genetic and/or medical conditions mimicking ADHD symptoms;
   * treatment with psychotropic medications other than ADHD medications.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We enrolled 67 individuals with ADHD and 70 typically developing youths (TDY) aged between 4 and 16 years. Individuals with ADHD were recruited from the Child and Adolescent Neuropsychiatry Unit, University of Sassari, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
To examine the association of ADHD with temperament dimensions and low cortisol levels, building on previous research that these may represent potential markers of low behaviour inhibition and under-arousal in the disorder. | six months
  Specifically:
  * we first investigate whether temperament dimensions and awakening cortisol level differ between youths with ADHD and controls and correlate with ADHD symptoms (inattention and hyperactivity-impulsivity).
  * Second, we examine whether the three temperament dimensions are associated with awakening cortisol levels.
To evaluate the association between cortisol levels and co-morbidity severity symptoms. | six months
  We test the association of oppositional-defiant and anxiety traits with the temperament dimensions and cortisol levels, and whether the association of ADHD with each temperament or cortisol measure remains when controlling for these comorbid psychiatric traits.

CONTACTS AND LOCATIONS:
Overall Officials: ALESSANDRA CARTA, Principal Investigator — Sassari University
Locations (2):
- Italy (2):
  - Alessandra Carta, Sassari
  - Complex Operating Unit of Child and Adolescent Neuropsychiatry - University of Sassari, Sassari

IPD SHARING:
Plan to Share IPD: No
Statistical Analyses were performed using the software R (version R 3.4.1). Analysis of variance covaring for sex (ANCOVA) was used to compare the two groups on the three temperament dimensions and on the awakening cortisol levels. A series of linear regression model analyses were used to test the association of temperament dimensions and cortisol levels with ADHD traits and the oppositional-defiant and anxiety traits. To test the difference between cortisol levels on- and off- methylphenidate treatment in participants with ADHD, we performed repeated measures analysis of variance. Before analysis, cortisol levels were log-transformed to normal. Analyses were then carried out using standardized scores for all measures.

REFERENCES:
- [Background] Karalunas SL, Fair D, Musser ED, Aykes K, Iyer SP, Nigg JT. Subtyping attention-deficit/hyperactivity disorder using temperament dimensions: toward biologically based nosologic criteria. JAMA Psychiatry. 2014 Sep;71(9):1015-24. doi: 10.1001/jamapsychiatry.2014.763. PMID 25006969
- [Result] Karalunas SL, Fair D, Musser ED, Aykes K, Iyer SP, Nigg JT. Notice of Retraction and Replacement. Karalunas et al. Subtyping attention-deficit/hyperactivity disorder using temperament dimensions: toward biologically based nosologic criteria. JAMA Psychiatry. 2014;71(9):1015-1024. JAMA Psychiatry. 2018 Apr 1;75(4):408-409. doi: 10.1001/jamapsychiatry.2018.0013. No abstract available. PMID 29516086
- [Result] Isaksson J, Nilsson KW, Nyberg F, Hogmark A, Lindblad F. Cortisol levels in children with attention-deficit/hyperactivity disorder. J Psychiatr Res. 2012 Nov;46(11):1398-405. doi: 10.1016/j.jpsychires.2012.08.021. Epub 2012 Sep 10. PMID 22974590